CLINICAL TRIAL: NCT07010354
Title: An International, Multi-centre Observational Study to Evaluate Safety, Performance, and Clinical Benefit of the BeFlow Iliac Covered Stent System
Brief Title: An Observational Study to Evaluate Safety, Performance, and Clinical Benefit of BeFlow
Status: Recruiting | Type: Observational
Sponsor: Bentley InnoMed GmbH (Industry)
Collaborators: ID3 Medical (Other)
Responsible Party: Sponsor
Other Study IDs: PM15-01 BeFlow
Record Dates: First submitted 2025-05-28; First posted 2025-06-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Iliac Artery Stenosis; Iliac Artery Occlusion
MeSH Terms: interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stenting — Endovascular treatment of stenosed or occluded iliac arteries: Permanent intraluminal placement of a covered stent

SUMMARY:
This international, observational multi-centre study of the device BFI will monitor technical success of the implantation, data regarding clinical performance, clinical benefit, as well as potential unknown side effects pursuant to the Intended Purpose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for permanent intraluminal placement in iliac arteries for restoring and improving the patency impaired by arteriosclerosis or other stenoses that may be treated by stenting according to the IFU of the BFI
* Patient is capable and willing to sign an informed consent
* Patients ≥18 years of age at the time of consent

Exclusion Criteria:

* Patients with any contraindication according to the IFU
* Previous stenting of the target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) suffering from stenotic lesions in the iliac arteries caused by arteriosclerosis or other pathologies that may be treated by stenting.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 12 months

SECONDARY OUTCOMES:
Rate of covered stent-related complications | 1 month and 12 months
Rate of technical success | up to 1 month
  successful positioning and deployment of the stents
Primary patency rate | up to 60 months
Secondary patency rate | up to 60 months
Primary assisted patency rate | up to 60 months
Change of Rutherford Classification | up to 60 months
Change of ABI | up to 60 months
Freedom from TLR | up to 60 months
Freedom from MACE | up to 60 months

CONTACTS AND LOCATIONS:
Locations (2):
- AZ Sint Blasius, Dendermonde, Belgium
- EOC - Ente Ospedaliero Cantonale, Lugano, Canton Ticino, Switzerland